CLINICAL TRIAL: NCT00349934
Title: IMP321 Phase I Study in Metastatic Breast Carcinoma Patients Receiving First-line Paclitaxel
Brief Title: IMP321 Plus First-line Paclitaxel in Metastatic Breast Carcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Immutep S.A.S. (Industry)
Collaborators: Umanis (Industry)
Responsible Party: F. Triebel, Chief Medical Officer, Immutep S.A.
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P005; Umanis-CRO0425
Record Dates: First submitted 2006-07-07; First posted 2006-07-10 (Estimated); Last update posted 2010-01-07 (Estimated); Status verified 2010-01

CONDITIONS: Metastatic Breast Cancer
Keywords: Metastatic breast cancer; IMP321; hLAG-3Ig; LAG-3; CD223; Chemotherapy; Paclitaxel; Combination therapy
MeSH Terms: conditions — Breast Neoplasms | interventions — soluble LAG-3 protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): IMP321
  Interventions: Biological: IMP321

INTERVENTIONS:
Biological: IMP321 — This study is an open label, non-randomized, fixed dose-escalation phase I study, performed in ambulatory setting with patients receiving as a first line chemotherapy for metastatic breast carcinoma the standard 6 cycles of paclitaxel (80 mg/m² at D1, D8 and D15 of every 4-week cycle).
  Three IMP321 dose levels (250 µg, 1,250 µg and 6,250 µg) will be evaluated in three cohorts of 8 patients. At any given dose level the patients will be administered one dose every two weeks for a total of 24 weeks (12 s.c. injections in total), separated by 13-day intervals free of IMP321 administration.
  The repeated single doses will be administered on D2 and D16 of the 4-week cycles, on the day which follows chemotherapy.
  Other Names: LAG-3; hLAG-3Ig; CD223

SUMMARY:
Open label, non-randomized, fixed dose-escalation phase I study, performed in ambulatory setting in patients receiving as a first line chemotherapy for metastatic breast carcinoma the standard 6 cycles of weekly paclitaxel (80 mg/m² at D1, D8 and D15 of a 4-week cycle). Three IMP321 doses (0.25, 1.25 and 6.25 mg) will be tested and given at D2 and D16 of this 4-week cycle, for 6 courses.

DETAILED DESCRIPTION:
This study is an open label, non-randomized, fixed dose-escalation phase I study, performed in ambulatory setting with patients receiving as a first line chemotherapy for metastatic breast carcinoma the standard 6 cycles of paclitaxel (80 mg/m² at D1, D8 and D15 of every 4-week cycle). Twenty mg i.v. dexamethasone will be given in the first cycle before each paclitaxel infusion. Corticosteroids will not be administered after the first chemotherapy cycle if the first 3 i.v. infusions of paclitaxel have been well tolerated.

Three IMP321 dose levels (0.25, 1.25 and 6.25 mg) will be evaluated in three cohorts of at lesat 8 patients. At any given dose level the patients will be administered one dose every two weeks for a total of 24 weeks (12 injections in total), separated by 13-day intervals free of IMP321 administration.

The study drug will be given by subcutaneous injection:

* Cohort A: 0.25 mg s.c.
* Cohort B: 1.25 mg s.c.
* Cohort C: 6.25 mg s.c.

The repeated single doses will be administered on D2 and D16 of the 4-week cycles, on the day which follows chemotherapy.

After a screening performed between Week -2 and Day 1, patients will enter the main study period. Upon having completed the 6 cycles of IMP321 treatment at Week 23, they will have an ambulatory 'post-study' examination (at Week 25).

Cohort B will be undertaken once the safety and tolerability results of Cohort A have been satisfactory; the investigator will take his decision for involving the last 8 patients of the study after the 6th administration (Week 13 assessment) of the fifth patient of Cohort A. All cohorts will follow the same schedule

Standard clinical and laboratory safety examinations, CT scan and pharmacodynamic (PD) blood tests will be performed. A complete examination will be carried out at Week 13 (after the 6th drug dosing) and Week 25.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stage IV breast adenocarcinoma, histologically proven by biopsy of the primary tumor and/or a metastasis.
* Female not pregnant (or with negative pregnancy test) or male.
* Fertile patients must use effective contraception during and for 3 months after drug administration.
* 18 years or above.
* ECOG performance status 0-1.
* Expected survival longer than three months.
* Resolution of toxicity of prior therapy to grade < 2 (except alopecia).
* With or without prior adjuvant or neoadjuvant chemotherapy (authorized).
* With or without hormone therapy in adjuvant and/or the advanced setting (authorized).
* Evidence of measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST).
* Biphosphonate therapy must have started at least 4 weeks prior to first dosing of the study drug.
* Asthma or chronic obstructive pulmonary disease allowed provided daily systemic corticosteroid therapy is not required.
* Total white cell count ≥ 3.109/L.
* Platelet count ≥ 100.109/L.
* Hemoglobin > 9 g/dL or > 5.58 mmol/L.
* Serum creatinine < 160 µmol/L.
* Total bilirubin < 20 mmol/L, except for familial cholemia (Gilbert's disease).
* Serum ASAT and ALAT < 3 times the upper limit of normal or < 5 times upper limit of normal if liver metastases are present.
* Able to give written informed consent and to comply with the protocol.

Exclusion Criteria:

* Prior chemotherapy for metastatic breast adenocarcinoma.
* Disease-free interval < 12 months from last dose of adjuvant chemotherapy.
* Prior high-dose chemotherapy requiring hematopoietic stem cell rescue.
* Inflammatory carcinoma.
* Systemic chemotherapy, hormone or endocrine therapy given as breast cancer therapy within 30 days prior to first dosing of the study drug.
* Any investigational drug within 30 days prior to first dosing of the study drug.
* Candidate for treatment with trastuzumab or administration of trastuzumab within 30 days prior to first dosing of the study drug.
* Known cerebral or leptomeningeal metastases.
* Pregnancy or breast feeding.
* Serious intercurrent infection within the 30 days prior to first dosing of the study drug.
* Motor or sensory peripheral neuropathy ≥ 2 according to the National Cancer Institute criteria.
* Congestive heart failure.
* Active acute or chronic infection.
* Active autoimmune disease requiring immunosuppressive therapy.
* Known HIV positivity.
* Life threatening illness unrelated to cancer.
* Previous malignancies within the last two years other than breast carcinoma, successfully treated squamous cell carcinoma of the skin or in situ carcinoma of the cervix treated with cone biopsy.
* Previous history of major psychiatric disorder requiring hospitalization or any current psychiatric disorder that would impede the patient's ability to provide informed consent or to comply with the protocol.
* Corticosteroids unless used as substitutive therapy or before each injection of paclitaxel.
* Past history of severe allergic episodes and/or Quincke edema.
* Past or present history of any organic disorder likely to modify absorption, distribution or elimination of the study drug.
* Alcohol or substance abuse disorder.
* Radiotherapy within the 30 days prior to first dosing of the study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2006-07; Primary Completion 2009-11 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Evaluate clinical and laboratory safety and tolerability profiles | 6 months
Determine pharmacodynamic parameters | 6 months

SECONDARY OUTCOMES:
Objective response rate (OR) using RECIST criteria | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Maya Gutierrez, M.D, Principal Investigator — Centre René Huguenin
Locations (3):
- France (3):
  - Hôpital Européen Georges Pompidou, Paris
  - Hôpital Tenon, Paris
  - Centre René Huguenin, Saint-Cloud

REFERENCES:
- [Derived] Brignone C, Gutierrez M, Mefti F, Brain E, Jarcau R, Cvitkovic F, Bousetta N, Medioni J, Gligorov J, Grygar C, Marcu M, Triebel F. First-line chemoimmunotherapy in metastatic breast carcinoma: combination of paclitaxel and IMP321 (LAG-3Ig) enhances immune responses and antitumor activity. J Transl Med. 2010 Jul 23;8:71. doi: 10.1186/1479-5876-8-71. PMID 20653948
- See also: Sponsor's website — http://www.immutep.com